CLINICAL TRIAL: NCT04739865
Title: The Safety and Efficacy Of Psilocybin as an Adjunctive Therapy in Participants With Treatment Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: COMPASS Pathways (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COMP003
Record Dates: First submitted 2020-09-22; First posted 2021-02-05 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 25 mg COMP360 Psilocybin (Experimental): 25 mg COMP360 Psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Open label
  Other Names: COMP360

SUMMARY:
The Safety and Efficacy of Psilocybin as an Adjunctive Therapy in Participants with Treatment-Resistant Depression

DETAILED DESCRIPTION:
A recent open label study of the effects of psilocybin in participants with treatment-resistant depression (TRD) showed rapid significant decrease of depressive symptoms after treatment with psilocybin coupled with psychological support. Over 40% of participants sustained response at 3 months. In this study, the aim is to explore effectiveness of 25 mg of psilocybin as an adjunctive therapy in participants with TRD.

ELIGIBILITY:
Inclusion Criteria:

1. Signed ICF.
2. 18 years of age or older
3. At least moderate MDD
4. Hamilton Depression Rating Scale (17 item) score ≥18
5. Currently receiving treatment with a selective serotonin reuptake inhibitor
6. Failure to respond to an adequate dose and duration of 2, 3, or 4 pharmacological treatments
7. McLean Screening Instrument for Borderline Personality Disorder <7 at Screening (V1).
8. Ability to complete all protocol required assessment tools without any assistance or alteration to the copyrighted assessments, and to comply with all study visits.

Exclusion Criteria:

Psychiatric Exclusion Criteria:

1. Current or past history of schizophrenia, psychotic disorder (unless substance induced or due to a medical condition), bipolar disorder, delusional disorder, paranoid personality disorder, schizoaffective disorder, or borderline personality disorder, as assessed by medical history, McLean Screening Instrument for Borderline Personality Disorder and a structured clinical interview (version 7.0.2 MINI).
2. Prior electroconvulsive therapy and/or ketamine for current episode.
3. Ongoing use of an antidepressant medication, including augmentation or combination therapies, other than a single SSRI
4. Current psychological therapies that will not remain stable within 21 days of the psilocybin session. Psychological therapies cannot be initiated within 21 days of baseline.
5. Current (within the last year) alcohol or substance use disorder as informed by DSM 5 (diagnosed by MINI 7.0.2) at Screening (V1).
6. Significant suicide risk as defined C-SSRS within the past year
7. Depression secondary to other severe medical conditions according to clinicians' judgement.
8. Other personal circumstances and behaviour judged to be incompatible with establishment of rapport or safe exposure to psilocybin, including exposure to psilocybin within the past year and use of psychedelics, such as ayahuasca, during the current depressive episode.

   General Medical Exclusion Criteria:
9. Women who are pregnant, nursing or planning a pregnancy.
10. Cardiovascular conditions
11. Uncontrolled or insulin dependent diabetes.
12. Seizure disorder.
13. Positive urine drug screen for illicit drugs or drugs of abuse
14. Current enrolment in any investigational drug or device study or participation in such within 30 days prior to Screening (V1).
15. Current enrolment in another clinical study of an investigational medical or participation in such within 30 days of Screening (V1).
16. Abnormal and clinically significant results on the physical examination, vital signs, ECG or laboratory tests at Screening (V1).
17. Any other clinically significant cardiovascular, pulmonary, gastrointestinal, hepatic, renal or any other major concurrent illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if he/she takes part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Goodwin, Principal Investigator — University of Oxford
Locations (2):
- Kadima Neuropsychiatry Institute, La Jolla, California, United States
- Sheaf House, Tallaght Hospital, Dublin, Ireland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient first visit: 10 August 2020 Last patient last visit: 13 October 2021
Period: Overall Study
Arm/Group | 25 mg COMP360 Psilocybin
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Psilocybin: 25mg Psilocybin
  Psilocybin: Open label
Arm/Group | Psilocybin
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (10.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 9
  Ireland | 10

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Depressive Symptoms
Description: Change in Montgomery-Asberg Depression Rating Scale (MADRS) total score from Baseline to 3 weeks post psilocybin administration.
  The minimum and maximum MADRS total score values are 0 and 60 and a higher score means a worse outcome.
Time Frame: 3 weeks
Population: Full analysis set - all participants who receive study drug and have at least 1 post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 25 mg COMP360 Psilocybin
Number analyzed (Participants) | 19
units on a scale | -14.9 (11.97)

2. Secondary Outcome: Incidence of Response
Description: The proportion of participants with a response (defined as a ≥ 50% improvement in Montgomery-Asberg Depression Rating Scale [MADRS] total score from Baseline) at Week 3 post psilocybin administration.
  The minimum and maximum MADRS total score values are 0 and 60 and a higher score means a worse outcome.
Time Frame: 3 weeks
Population: Full analysis set - all participants who receive study drug and have at least 1 post-baseline efficacy assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mg COMP360 Psilocybin
Number analyzed (Participants) | 19
Participants | 8

3. Secondary Outcome: Incidence of Remission
Description: The proportion of participants with remission (defined as Montgomery-Asberg Depression Rating Scale [MADRS] total score ≤ 10) at Week 3 post psilocybin administration The minimum and maximum MADRS total score values are 0 and 60 and a higher score means a worse outcome.
Time Frame: 3 weeks
Population: Full analysis set - All participants who receive study drug and have at least 1 post-baseline efficacy assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mg COMP360 Psilocybin
Number analyzed (Participants) | 19
Participants | 8

4. Secondary Outcome: Improvement in Clinical Global Impression - Severity
Description: Changes from Baseline in Clinical Global Impression-Severity score at Week 3 post psilocybin administration.
  The minimum and maximum values are 1 and 7 and a higher score means a worse outcome.
Time Frame: 3 weeks
Population: Full analysis set - All participants who receive study drug and have at least 1 post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 25 mg COMP360 Psilocybin
Number analyzed (Participants) | 19
units on a scale | -1.3 (1.29)

ADVERSE EVENTS:
Time Frame: Up to 3 weeks
Description: Safety analysis set - All participants who receive study drug.
Arm/Group | 25 mg COMP360 Psilocybin
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 12/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mg COMP360 Psilocybin (N=19)
Palpitations (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1)
Blood Pressure Increased (Investigations) | 3 (3)
Headache (Nervous system disorders) | 6 (6)
Dizziness (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT04739865/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT04739865/SAP_001.pdf